CLINICAL TRIAL: NCT05067049
Title: Evaluation of the Impact of a Connected Application on the Follow-up of Patients Treated for Glial Lesions Operated: a Prospective, Randomized Study
Brief Title: Evaluation of the Impact of a Connected Application on the Follow-up of Patients Treated for Glial Lesions Operated
Acronym: TELEGLIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Clairval Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A03009-46
Record Dates: First submitted 2021-09-10; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Quality of Life; Phone Use, Cell; Glial Scar
MeSH Terms: conditions — Cell Phone Use; Gliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connected EORTC-C30 arm (quality of life questionnaires on pad, phone,...) (Experimental): The patients in this arm will have connected mobile app at home and they will regularly fill questionnaires. There are two different questionnaires : one with 14 questions about patient's quality of life and about the evolution of his surgical scar. One with 9 questions only about quality of life. They will also have meetings with physicians.
  Interventions: Device: Connected application arm
- No QoL online follow-up arm (Other): The patient haven't any questionnaires to fill at home. This is the normal management of the pathology. They only have different meeting with the specialist,as usual.
  Interventions: Device: Unconnected arm

INTERVENTIONS:
Device: Connected application arm — patients have to respond different questionnaires about their quality of life on the mobile app.
  And follow-up visits with the physicians as usual
  Arms: Connected EORTC-C30 arm (quality of life questionnaires on pad, phone,...)
Device: Unconnected arm — Follow-up visits with the pysicians as usual
  Arms: No QoL online follow-up arm

SUMMARY:
This study is to evaluate the efficacy of a mobile app for monitoring the quality of life of patients but also on detection delay of side effects and/or complications linked to the therapeutic management. This allow to adapt their care more quickly, through a prospective randomized study. The impact of this connected monitoring of patients' anxiety will also be evaluated in this study as well as the time taken by the medical team to manage alerts generated by this application.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old without upper age limit.
* Subject operated for a non-recurrent glioma (grade II or III or IV glioma / glioblastoma) according to the WHO classification 2016;
* Subject with a connected support (smartphone,...) to download the connected tracking application.
* Unprotected adult within the meaning of the law
* Subject affiliated to a health insurance scheme
* Subject having signed an informed written consent

Exclusion Criteria:

* Minor subject, pregnant or breastfeeding woman;
* Subject under a measure of legal protection, guardianship or deprived of liberty by judicial or administrative decision;
* Antipsychotic treatment (neuroleptic or lithium)
* Subjects with documented cognitive disorders (Alzheimer, other dementia)
* Subject with a personal medical history of psychiatry
* Subject unable to complete a questionnaire on his own (inability to read French language , severe cognitive disorders)
* Medical contraindication to performing an MRI (pace-maker) or scanner;
* Subject refusing to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of the impact of the connected mobile monitoring application on the quality of life, at 6 months, of patients treated for an operated glioma. | 6 months
  The primary outcome measure is the difference in quality of life assessed by the QLQ-BN20 scale at 6 months, compared to inclusion. This scale is made up of 20 items which are grouped into 4 dimensions (future uncertainty, visual disorder, motor dysfunction, and communication deficit) and 7 isolated items.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique privée, Marseille, France